CLINICAL TRIAL: NCT06644807
Title: Neuromodulation Methods for Suppressing Phantom Limb Pain
Brief Title: Study of Phantom Limb Pain Suppression Using Neuromodulation Methods
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Skolkovo Institute of Science and Technology (Other)
Collaborators: Motorica LLC (Unknown); Federal center of brain research and neurotechnologies (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Skoltech-CNBR4
Record Dates: First submitted 2024-09-02; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Phantom Limb Pain
Keywords: Neuromodulation; Phantom limb pain; Neuropathic pain; Neurostimulation; Chronic pain; Peripheral nerve stimulation; PNS; Spinal cord stimulation; SCS; Dorsal root ganglion stimulation; DRG; Cortical stimulation; Amputation; Amputees; Upper-limb injury
MeSH Terms: conditions — Phantom Limb; Neuralgia; Chronic Pain; Arm Injuries | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Peripheral nerve stimulation (Experimental)
  Interventions: Procedure: Peripheral Nerve Stimulation
- Spinal cord stimulation (Experimental)
  Interventions: Procedure: Spinal cord stimulation
- Motor Cortex Stimulation (Experimental)
  Interventions: Procedure: Motor Cortex Stimulation
- Dorsal Root Ganglion Stimulation (Experimental)
  Interventions: Procedure: Dorsal Root Ganglion Stimulation

INTERVENTIONS:
Procedure: Motor Cortex Stimulation — Motor Cortex Stimulation (MCS) is a neuromodulation technique that involves the surgical implantation of electrodes over the motor cortex, typically targeting the precentral gyrus, to deliver electrical stimulation. The procedure involves placing an electrode grid or strip on the dura mater overlying the motor cortex, which is identified via neuroimaging techniques such as functional MRI or neuronavigation. Once implanted, the electrodes are connected to an implanted pulse generator (IPG), which delivers adjustable electrical impulses.
  Arms: Motor Cortex Stimulation
Procedure: Spinal cord stimulation — Spinal Cord Stimulation (SCS) is a neuromodulation that involves the implantation of a device that delivers electrical impulses to the spinal cord through an electrode placed in the epidural space. The stimulation alters pain signals before they reach the brain, effectively masking or reducing the sensation of pain.
  Arms: Spinal cord stimulation
Procedure: Peripheral Nerve Stimulation — Peripheral Nerve Stimulation (PNS) is a neuromodulation technique used to treat chronic pain. The procedure starts with a preoperative assessment, including imaging to identify the target peripheral nerve. Under local anesthesia, a thin, insulated electrode is implanted near the nerve, usually with the help of fluoroscopic or ultrasound guidance for precision.
  Arms: Peripheral nerve stimulation
Procedure: Dorsal Root Ganglion Stimulation — Dorsal Root Ganglion Stimulation (DRGS) is a targeted neuromodulation technique for managing chronic pain. The procedure begins with a thorough preoperative assessment, including imaging to locate the specific dorsal root ganglion (DRG) associated with the pain. Under local anesthesia, a small electrode is implanted near the DRG. This is done through a minimally invasive procedure, often guided by fluoroscopy or CT imaging to ensure precise placement.
  Arms: Dorsal Root Ganglion Stimulation

SUMMARY:
This study assesses the effectiveness of neuromodulation in alleviating pain through the stimulation of peripheral nerves. The research involves implanting electrodes for test stimulation of peripheral nerves (PNS - Peripheral Nerve Stimulation), spinal cord (SCS - Spinal Cord Stimulation), dorsal root ganglia (DRGS - Dorsal Root Ganglion Stimulation), and motor cortex (MCS - Motor Cortex Stimulation). The study aims to explore the use of neuromodulation for pain relief in patients experiencing pain due to upper or lower limb amputation.

ELIGIBILITY:
Inclusion Criteria:

* Amputation of the upper limb at the level of the forearm or upper arm, or amputation of the lower limb at the level of the lower leg or thigh.
* Age between 18 and 65 years.
* Duration since amputation is at least 6 months.
* Presence of persistent chronic pain syndrome rated between 4 and 10 on the Visual Analog Scale (VAS).
* Absence of pregnancy at the time of implantation, confirmed by a pregnancy test (for female participants only).
* Signed consent to participate in the study.

Exclusion Criteria:

* Presence of severe somatic pathology that hinders surgical treatment and participation in the study.
* Presence of psychiatric disorders (including a history of), severe depression, suicidal tendencies, or a history of suicide attempts.
* Presence of severe orthopedic deformity in the limb above the level of amputation.
* History of cancer.
* History of epilepsy.
* Complicated traumatic brain injury (TBI) or a history of stroke.
* Inability to undergo electrostimulation due to other somatic pathology.
* Purulent-septic pathology.
* Drug addiction (including a history of).
* Congenital anomaly of upper limb development.
* Anomalies in the development of the central and peripheral nervous systems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | Up to 4 months
  The Visual Analog Scale (VAS) is a 10 cm line used to measure pain intensity. One end of the line represents "no pain," while the other end signifies "worst possible pain." The line can be either horizontal or vertical.
SF-36 | up to 1 year
  The questionnaire consists of 36 items grouped into eight scales: physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, emotional well-being, and mental health. Each scale ranges from 0 to 100, where 100 represents full health. Higher scores indicate better quality of life, with two summary measures: physical and mental well-being.

SECONDARY OUTCOMES:
Sensory mapping | up to 4 months
  The sensory mapping procedure involved evoking sensations in phantom hands through peripheral nerve stimulation (PNS). Electrode pairs were selected, and stimulation parameters, with fixed pulse width and frequency were applied. Stimulation amplitude was gradually increased in 0.1-mA steps until participants rated their sensation intensity from 0 (no sensation) to 10 (uncomfortably intense). Upon reaching a score of 5, participants marked sensation location on a hand image and described the sensation's naturalness and intensity.
Pain detect | Up 1 year
  The questionnaire is intended for completion by a physician and combines a pain distribution diagram with a visual analog scale (VAS) and a section focused on identifying spontaneous and triggered neuropathic pain symptoms. It also assesses the nature of pain using the diagram, categorizing it as constant, episodic, or constant with episodes, among others. The questionnaire comprehensively reflects all possible pain parameters, allowing for clear tracking of pain dynamics over time. Its diagnostic accuracy is 83%.
DN 4 | up to 1 year
  The DN4 (Douleur Neuropathique 4) questionnaire is a diagnostic tool designed to identify neuropathic pain, caused by nerve damage. It includes 10 items divided into two sections. The first part consists of seven questions that assess the patient's pain symptoms, such as burning, tingling, electric shocks, or numbness. The second part involves a clinical examination where the physician tests for reduced sensitivity to touch and pinprick, as well as pain response to light brushing. Each item is scored with 1 point for "Yes" and 0 for "No." A total score of 4 or higher indicates a high probability of neuropathic pain.
Hospital Anxiety and Depression Scale, HADS | up to 1 year
  The Hospital Anxiety and Depression Scale (HADS) is a widely used screening tool designed to assess anxiety and depression levels in patients in non-psychiatric hospital settings. It consists of 14 items, divided into two subscales: seven questions assess anxiety (HADS-A) and seven assess depression (HADS-D). The items focus on emotional and cognitive symptoms rather than physical symptoms, making it suitable for patients with medical conditions. Each item is scored on a scale of 0 to 3, with total scores for each subscale ranging from 0 to 21. A score of 8 or more on either subscale suggests the presence of anxiety or depression. The HADS is valued for its simplicity and reliability in clinical and research settings.
Sensory threshold | up to 6 months
  In this experiment, the goal is to determine the minimum stimulation amplitude that elicits a sensory response. Participants are shown the numbers 1 and 2 on a screen, with stimulation activated simultaneously upon the appearance of one of the numbers. Their task is to identify when the stimulation occurred and input their answer on a keyboard. An expanded version of the experiment may provide stimulation during both moments, requiring participants to determine which moment had a higher stimulation level. The results will yield a psychophysical curve that illustrates the relationship between response accuracy and stimulation amplitude, as well as the participants' ability to differentiate stimulation parameters. It is anticipated that over time, the sensory threshold will shift, leading to increased accuracy in parameter identification.

OTHER OUTCOMES:
OPUS | up to 4 months
  OPUS (Optimal Patient Utilization System) is a clinical decision support tool designed to enhance patient care through improved resource management and treatment efficiency. It utilizes advanced algorithms and data analytics to optimize patient scheduling, treatment pathways, and staff allocation within healthcare facilities. By analyzing patient demographics, medical history, and treatment outcomes, OPUS helps clinicians make informed decisions about resource allocation and care delivery. The system aims to reduce wait times, streamline operations, and improve overall patient satisfaction. Additionally, OPUS provides real-time feedback and reporting capabilities, enabling healthcare providers to monitor performance metrics and identify areas for improvement, ultimately enhancing the quality of care.
PEQ (Prosthesis Evaluation Questionnaire) | up to 4 months
  The Prosthesis Evaluation Questionnaire (PEQ) is a standardized assessment tool designed to evaluate the functional and psychosocial outcomes of individuals using prosthetic devices. Comprising various domains, the PEQ addresses aspects such as mobility, activity level, and quality of life, allowing users to report their experiences and satisfaction with their prosthesis. The questionnaire includes specific items that gauge the user's perception of their prosthetic limb's comfort, functionality, and impact on daily activities. By providing a comprehensive view of the user's experience, the PEQ helps healthcare professionals identify areas for improvement in prosthetic design and rehabilitation strategies. The results from the PEQ can inform clinical decisions and enhance personalized care, ultimately leading to better patient outcomes and satisfaction.

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Federal Center of Brain Research and Neurotechnologies of the Federal Medical Biological Agency of Russia, Moscow, Moscow
  - Federal Center of Brain Research and Neurotechnologies of the Federal Medical Biological Agency of Russia, Moscow